CLINICAL TRIAL: NCT03037372
Title: Statin Adjunct Therapy Among HAART-treated Adults in Sub-Saharan Africa: Equivalence of Atorvastatin and Rosuvastatin
Brief Title: Statin Adjunct Therapy Among ART-treated Adults in Sub-Saharan Africa: Atorvastatin and Rosuvastatin Equivalence Trial
Acronym: STAR
Status: Unknown | Phase: Phase 3 | Type: Interventional
Last Known Status: Not yet recruiting
Sponsor: Makerere University (Other)
Collaborators: University of Oxford (Other); Case Western Reserve University (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: DN2017
Record Dates: First submitted 2017-01-10; First posted 2017-01-31 (Estimated); Last update posted 2017-01-31 (Estimated); Status verified 2017-01

CONDITIONS: HIV Infection
Keywords: adults; antiretroviral therapy
MeSH Terms: conditions — HIV Infections | interventions — Atorvastatin; Rosuvastatin Calcium

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (4):
- ART-Atorvastatin adjunct therapy (Experimental): ART, atorvastatin
  Interventions: Drug: ART, Atorvastatin
- ART-Rosuvastatin adjunct therapy (Experimental): ART, rosuvastatin
  Interventions: Drug: ART, Rosuvastatin
- ART-without statin adjunct therapy (Experimental): ART, no statin
  Interventions: Drug: ART, No statin
- Healthy-HIV-negative (Experimental): Age-matched HIV-negative, healthy volunteers from the same community
  Interventions: Drug: Healthy-HIV-negative

INTERVENTIONS:
Drug: ART, Atorvastatin — ART, Atorvastatin
  Other Names: Atovastatin adjunct therapy
  Arms: ART-Atorvastatin adjunct therapy
Drug: ART, Rosuvastatin — ART, Rosuvastatin
  Other Names: Rosuvastatin adjunct therapy
  Arms: ART-Rosuvastatin adjunct therapy
Drug: ART, No statin — ART, No statin
  Other Names: No statin adjunct therapy
  Arms: ART-without statin adjunct therapy
Drug: Healthy-HIV-negative — Age-matched, Healthy HIV-negative
  Other Names: HIV-negative controls
  Arms: Healthy-HIV-negative

SUMMARY:
This study will determine whether 36 months of daily atorvastatin or rosuvastatin have equivalent effects in reduction of immune activation, inflammation and immune aging, when given as adjunct therapy among patients receiving antiretroviral therapy in an African cohort

DETAILED DESCRIPTION:
This is a randomized, open-label trial

ELIGIBILITY:
Inclusion Criteria:

* HIV-positive individuals 18 years and older, that have initiated three first-line drug highly active antiretroviral therapy within three months within the Infectious Diseases Institute HIV treatment cohort
* Individuals that provide written informed consent to participate in the clinical trial

Exclusion Criteria:

Individuals with dyslipidemia and eligible to receive or already receiving statin therapy

* Pregnant or lactating mothers
* Individuals with another active or controlled inflammatory condition
* Individuals with deranged liver function tests 3 fold and above

Ages: 18 Years to 90 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 320 (Estimated)
Dates: Start 2017-06-01 (Estimated); Primary Completion 2022-06-30 (Estimated); Study Completion 2022-12-31 (Estimated)

PRIMARY OUTCOMES:
Similar rate of reduction of immune activation between atorvastatin and rosuvastatin arms (p<o.05) | 12 months
  measured by percentage of HLADR+CD38+T-cells

SECONDARY OUTCOMES:
Similar rate of change of immune aging markers, between ART-treated adults with and without statin (atorvastatin and rosuvastatin) adjunct therapy arms (P-value<0.05) | 36 months
  Measured by Percentage of CD4+ and CD8+ naive T-cells or percentage of expressing Ki67 T-cells or percentage of low CFSE+T-cells or increase in percentage of CD28-/CD57+ T-cells or percentage of individuals with low host responses to influenza vaccine among HIV-infected adults at ART initiation
Similar rate of reduction of inflammatory markers, between atorvastatin and rosuvastatin arms (p<0.05) | 36 months
  Measured by levels of IL6 in pg/ml, hsCRP in pg/ml, d-dimers in pg/ml, IFABP in pg/ml, and LPS in pg/ml
Biological pathways affected by atorvastatin and rosuvastatin | 36 months
  number of genes down-regulated by either atorvastatin or rosuvastatin

CONTACTS AND LOCATIONS:
Overall Officials: Damalie Nakanjako, PhD, Principal Investigator — Makerere University College of Health Sciences

IPD SHARING:
Plan to Share IPD: Yes
Data will be shared with the Infectious Diseases Institute, according to the IDI data sharing policy

REFERENCES:
- [Result] Funderburg NT, Jiang Y, Debanne SM, Labbato D, Juchnowski S, Ferrari B, Clagett B, Robinson J, Lederman MM, McComsey GA. Rosuvastatin reduces vascular inflammation and T-cell and monocyte activation in HIV-infected subjects on antiretroviral therapy. J Acquir Immune Defic Syndr. 2015 Apr 1;68(4):396-404. doi: 10.1097/QAI.0000000000000478. PMID 25514794
- [Result] Nakanjako D, Ssinabulya I, Nabatanzi R, Bayigga L, Kiragga A, Joloba M, Kaleebu P, Kambugu AD, Kamya MR, Sekaly R, Elliott A, Mayanja-Kizza H. Atorvastatin reduces T-cell activation and exhaustion among HIV-infected cART-treated suboptimal immune responders in Uganda: a randomised crossover placebo-controlled trial. Trop Med Int Health. 2015 Mar;20(3):380-90. doi: 10.1111/tmi.12442. Epub 2015 Jan 6. PMID 25441397